CLINICAL TRIAL: NCT02411487
Title: Meibomian Gland Dysfunction (MGD) and Tear Cytokines After Cataract Surgery According to Preoperative Meibomian Gland Status
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-1103
Record Dates: First submitted 2015-03-05; First posted 2015-04-08 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — TEAR
Oversight: Data Monitoring Committee: No

SUMMARY:
To investigate the possible mechanisms by which cataract surgery aggravates meibomian gland dysfunction (MGD), the investigators evaluated the changes in tear cytokines and ocular surface parameters after cataract surgery according to the preoperative MGD grade.

ELIGIBILITY:
Inclusion Criteria:

* males or non-pregnant females aged between 55 to 80 years-old.

Exclusion Criteria:

* had a history of ocular diseases, such as ocular infection, ocular allergy, and autoimmune disease, as well as patients with continuous use of topical ocular medications before surgery, or histories of ocular surgery or ocular injury.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 55 eyes from 55 patients who underwent cataract surgery were included.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2015-08-03 (Actual); Study Completion 2015-08-03 (Actual)

PRIMARY OUTCOMES:
inflammatory tear cytokine concentration | 1 month after cataract surgery
  comparison of tear cytokines (IL-2,4,10,17a, INF-r, TNF-a) concentrations in patients with or without newly diagnosed chronic GVHD after SCT using a multiplex immunobead assay
ocular surface staining | 1 month after cataract surgery
tear film break-up time, | 1 month after cataract surgery
conjunctival injection, | 1 month after cataract surgery
Schirmer's test I | 1 month after cataract surgery
ocular surface disease index | 1 month after cataract surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Li XM, Hu L, Hu J, Wang W. Investigation of dry eye disease and analysis of the pathogenic factors in patients after cataract surgery. Cornea. 2007 Oct;26(9 Suppl 1):S16-20. doi: 10.1097/ICO.0b013e31812f67ca. PMID 17881910
- [Background] Cyclin-dependent kinase inhibitory protein expression in human choroidal melanoma tumors. Mouriaux F,*(1) Maurage CA, Labalette P, Sablonniere B, Malecaze F, Darbon JM. Inv Ophthalmol Vis Sci 2000;41:2837-2843. Am J Ophthalmol. 2001 Jan;131(1):157. doi: 10.1016/s0002-9394(00)00922-3. No abstract available. PMID 11341889